CLINICAL TRIAL: NCT05818332
Title: Implementation of Routine Recording of Intraoperative Adverse Events According to ClassIntra® During the Sign-out Phase of the WHO Surgical Safety Checklist Using a Multifaceted, Tailored Implementation Strategy: Protocol of a Collaborative Before- and After-cohort Project
Brief Title: ClassIntra® for Better Outcomes in Surgery - CIBOSurg
Acronym: CIBOSurg
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2023-00330
Record Dates: First submitted 2023-03-15; First posted 2023-04-18 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Perioperative Patient Safety
Keywords: Perioperative safety; sign-out; intraoperative adverse events; ClassIntra®; hybrid design
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- before and after implementation cohort: consecutive cohort of 900 surgical patients (baseline)
  consecutive cohort of 900 surgical patients (after implementation with a multifaceted, tailored implementation strategy to improve adherence to the WHO SSC and routine recording of iAEs)
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention, observational only

SUMMARY:
Intra- and postoperative adverse events (iAEs and pAEs) occur in up to one third of all patients undergoing surgery. They are devastating to patients and costly to health care systems. Their number tends to increase due to the rising complexity of both the patient's risk profile and the surgical procedure. Postoperative deaths have been identified to be the third most frequent cause of death worldwide. Teamwork in surgery has been attributed to have a potentially great impact on avoiding postoperative morbidity. Up to 50% of all adverse in-hospital events were rated to be potentially preventable. However, their prevention typically requires a change in systems and individual behaviour. Standardised assessments of iAEs and pAEs are a prerequisite to develop and define strategies for prevention of AEs. While awareness of pAEs has highly risen through the introduction of the Clavien-Dindo classification, the most widely used classification for grading severity of pAEs, the relevance of transparent monitoring of iAEs is still highly undervalued.

ELIGIBILITY:
Inclusion Criteria:

- All in-hospital patients (consecutive or random sample) undergoing surgery from general surgery, vascular, surgery, orthopaedics/traumatology and urology in the operating room with anaesthesia involvement

Exclusion Criteria:

* Patients undergoing one-day-surgery (with or without anaesthesia-involvement)
* Procedures without anaesthesia-involvement (in- or out-patient)
* ASA risk classification (ASA) VI patients (brain-death, organ-donor)
* Follow-up procedure of a patient already included in the study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All in-hospital patients (consecutive) undergoing surgery in the operating room with anaesthesia involvement
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Intervention fidelity - component checklist completion | 2 months after the end of the implementation
  Checklist completion is defined as completeness of all ticks on the sign-out checklist taking into consideration the minimum standard.

SECONDARY OUTCOMES:
Intervention fidelity - component quality of checklist performance | Up to four months after the implementation
  Quality of the sign-out will be measured with the WHO behaviourally anchored rating scale (WHOBARS):
  Quality will be measured in a random sample of 20-25%, assessed in those centres with well-established sign-out in the baseline period and in all centres in the after-implementation phase.
Implementation fidelity - Quantitative and qualitative evaluation of critical implementation steps | Up to four months after the implementation
  Quantitative and qualitative evaluation of critical implementation steps followed or not (and why not) by each site, according to the proposed/designed implementation plan (template)
Intervention acceptability - extent of perception among stakeholders that the intervention is agreeable or satisfactory | Measured after the implementation
  Acceptability is the extent of perception among stakeholders that the intervention is agreeable or satisfactory. It will be measured according to the Acceptability of Intervention Measure (AIM).
Adaptation - extent to which sign-out and documentation of iAEs have been locally adapted | Checklist and process modifications classified according to FRAME.
  Adaptation is the extent to which sign-out and documentation of iAEs have been locally adapted. It will be measured by comparing the local checklists with the minimum standard sign-out.
Appropriateness - extent to which staff perceive the intervention as being a good fit, relevant and compatible with their setting | Measured after the implementation
  Appropriateness is the extent to which staff perceive the intervention as being a good fit, relevant and compatible with their setting. It will be measured by the Intervention Appropriateness Measure (IAM).
Feasibility - extent to which sign-out and documentation of iAEs can be successfully used or carried out within a given setting | Measured after the implementation
  Feasibility is the extent to which sign-out and documentation of iAEs can be successfully used or carried out within a given setting. It will be measured by the Feasibility of Intervention Measure FIM.
Sustainment | 12 months after the last patient out
  Sustainment is measured by comparing (full) adherence (defined as completeness of all ticks on the sign-out checklist) 12 months after implementation

OTHER OUTCOMES:
Qualitative conclusions | Longitudinal data collection before, during and after the implementation
  Qualitative conclusions about the effectiveness of the employed implementation strategy.
Characterising themes | Longitudinal data collection before, during and after the implementation
  Themes characterising the factors that influenced the observed implementation processes, based on the results from the contextual analysis.
Comprehensive Complication Index (CCI®) | Difference in CCI® before and after the implementation at hospital discharge and at 90 days after surgery
  CCI® (Comprehensive Complication Index) is the weighted sum of all pAEs according to Clavien-Dindo. It will be assessed at hospital discharge and at 90 days after surgery.
Severe iAEs according to ClassIntra® | Difference in number of severe iAEs before and after the implementation
  Severe iAEs according to ClassIntra® are defined as greater than or equal to grade III.
Total number of iAEs according to ClassIntra® | Difference in total number of iAEs before and after the implementation
  Total number of iAEs according to ClassIntra® occurring in the baseline and the after implementation period.
Severe pAEs according to Clavien-Dindo | Difference in number of severe iAEs before and after the implementation
  Severe pAEs according to Clavien-Dindo are defined as greater than or equal to grade IIIa. They will be assessed at hospital discharge and at 90 days after surgery.
Total number of pAEs according to Clavien-Dindo | Difference in total number of pAEs before and after the implementation
  Total number of pAEs according to Clavien-Dindo occurred in the baseline and the after implementation period. They will be assessed at hospital discharge and at 90 days after surgery.
Number of resulting actions due to the routine recording and discussion of iAEs during the sign-out | Difference in number of resulting actions before and after the implementation
  Resulting actions are e.g. preventive measures for anticipated pAEs.
Length of hospital stay | Difference in length of hospital stay before and after the implementation
  Length of hospital stay will be measured in days.

CONTACTS AND LOCATIONS:
Locations (10):
- Radboud UMC, Nijmegen, Netherlands
- Switzerland (9):
  - University Hospital Basel, Basel
  - Lindenhofspital, Bern
  - University Hospital Berne, Bern
  - Cantonal Hospital Graubünden, Chur
  - University Hospital Geneva, Geneva
  - University Hospital Lausanne, Lausanne
  - Cantonal Hospital Lucerne, Lucerne
  - Regional Hospital Lugano, Lugano
  - University Hospital Zurich, Zurich